CLINICAL TRIAL: NCT05043441
Title: A Ten-Week Online Acceptance and Commitment Therapy Intervention Guided by a Coach for Family Caregivers of People With Dementia: A Randomized Controlled Trial
Brief Title: A Ten-Week Online Acceptance and Commitment Therapy Intervention for Family Caregivers of People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Areum Han, Assistant professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AARG-21-846868
Record Dates: First submitted 2021-09-05; First posted 2021-09-14 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Depressive Symptoms
Keywords: Acceptance and Commitment Therapy; Alzheimer's Disease; Burden; Caregivers; Dementia; Mindfulness; Psychological health; Quality of life; Self-compassion; Stress; Depression; Anxiety; Guilt; Grief
MeSH Terms: conditions — Depression; Alzheimer Disease; Dementia; Psychological Well-Being; Anxiety Disorders | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and commitment therapy (ACT) group (Experimental): 10 weekly ACT sessions individually guided by a trained coach through Zoom videoconferencing with psychoeducation materials provided
  Interventions: Behavioral: Acceptance and commitment therapy (ACT)
- Psychoeducation control group (Sham Comparator): Care as usual with psychoeducation materials provided
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy (ACT) — Caregivers assigned to this intervention group will receive individual ACT sessions guided by a trained coach for one hour per week over 10 weeks through Zoom videoconferencing with psychoeducation materials provided.
  Arms: Acceptance and commitment therapy (ACT) group
Behavioral: Psychoeducation — The psychoeducation control group will receive care as usual with psychoeducation materials provided.
  Arms: Psychoeducation control group

SUMMARY:
This randomized controlled trial aims to assess the effects of a coach-guided ten-week videoconferencing acceptance and commitment therapy (ACT) program on mental health outcomes in depressed family caregivers of people with dementia (PwD) compared to the control group. A total of 32 family caregivers of PwD who meet the eligibility criteria will be recruited and randomized to either the intervention group or the control group. The hypotheses are that the ACT group will show improvements in depressive symptoms, other mental health outcomes, and ACT process measures at posttest and 3-month follow-up, compared to the control group.

DETAILED DESCRIPTION:
This randomized controlled trial aims to assess the effects of a coach-guided ten-week videoconferencing acceptance and commitment therapy (ACT) program on mental health outcomes in depressed family caregivers of people with dementia (PwD) compared to the control group. A total of 32 family caregivers of PwD who meet the eligibility criteria will be recruited and randomized to either the intervention group or the control group. Caregivers randomly assigned to the intervention group will receive individual ACT sessions guided by a trained coach for one hour per week over 10 weeks through Zoom videoconferencing with supplemental psychoeducation materials provided. Caregivers randomly assigned to the control group will receive care as usual with psychoeducation materials provided during the study period. Outcomes regarding caregivers' mental health and ACT processes will be collected at three time points (i.e., pretest, posttest, and 3-month follow-up) and compared between groups over time. The hypotheses are that the ACT group will show improvements in depressive symptoms, other mental health outcomes, and ACT process measures at posttest and 3-month follow-up, compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling adults (age 18 or over) who are currently taking the primary responsibility for the care of a relative with dementia living in the community
* having at least mild depression as measured by the Patient Health Questionnaire (PHQ)-9
* having a computer or a smartphone with the internet access at home and
* being able to provide informed consent

Exclusion Criteria:

* having cognitive, physical, or sensory deficits or language barriers (non-English communicator) that impede study participation
* having psychiatric hospitalizations or diagnoses of mental illness in the previous two years
* taking antipsychotic or anticonvulsant medication at the time of recruitment
* considering or planning to place family members of PwD in a nursing home within 6 months or
* having the possibility of study dropouts due to medical conditions of caregivers (e.g., surgery that may affect mental health) and their relatives with dementia (e.g., conditions that may impede study participation due to frequent hospitalization or death)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline to immediately after the intervention and 3 month follow-up on the Patient Health Questionnaire-9 | Change from baseline to immediately after the intervention and 3 month follow-up
  The Patient Health Questionnaire-9 is a 9-item questionnaire assessing depressive symptoms on a scale of 0 to 3. Scores range from 0 to 27. Higher scores indicate greater symptomatology in depression.

SECONDARY OUTCOMES:
Change from baseline to immediately after the intervention and 3 month follow-up on the Generalized Anxiety Disorder-7 | Change from baseline to immediately after the intervention and 3 month follow-up
  The Generalized Anxiety Disorder-7 is a 7-item questionnaire assessing anxiety on a scale of 0 to 3. Scores range from 0 to 21. Higher scores indicate greater anxiety.
Change from baseline to immediately after the intervention and 3 month follow-up on the Perceived Stress Scale | Change from baseline to immediately after the intervention and 3 month follow-up
  The Perceived Stress Scale is a 10-item questionnaire assessing stress on a scale of 0 to 4. Scores range from 0 to 40. Higher scores indicate greater stress.
Change from baseline to immediately after the intervention and 3 month follow-up on the World Health Organization Quality of Life - Psychological health component | Change from baseline to immediately after the intervention and 3 month follow-up
  World Health Organization Quality of Life - Psychological health component has 6 items measuring psychological quality of life on scale of 1 to 5. Scores range from 6 to 30. Higher scores denote higher quality of life in terms of psychological health.
Change from baseline to immediately after the intervention and 3 month follow-up on the Meuser Caregiver Grief Inventory | Change from baseline to immediately after the intervention and 3 month follow-up
  Marwit-Meuser Caregiver Grief Inventory Brief-Form is a 6-item self-report questionnaire assessing grief of caregivers on a scale of 1 to 5. Scores range from 6 to 30. Higher scores indicate higher levels of grief.
Change from baseline to immediately after the intervention and 3 month follow-up on the Caregiver Guilt Questionnaire | Change from baseline to immediately after the intervention and 3 month follow-up
  Caregiver Guilt Questionnaire is a 22-item self-report questionnaire assessing feelings of guilt in caregivers on a scale of 0 to 4. Scores range from 0 to 88. Higher scores indicate higher levels of guilt.
Change from baseline to immediately after the intervention and 3 month follow-up on the Self-Compassion Scale- Short Form | Change from baseline to immediately after the intervention and 3 month follow-up
  Self-Compassion Scale- Short Form is a 12-item self-report questionnaire assessing self-compassion on a scale of 1 to 5. Scores range from 12 to 60. Higher scores indicate higher levels of self-compassion.
Change from baseline to immediately after the intervention and 3 month follow-up on the Action and Acceptance Questionnaire-II | Change from baseline to immediately after the intervention and 3 month follow-up
  Action and Acceptance Questionnaire -II is a 7-item self-report questionnaire measuring psychological flexibility on a scale of 1 to 7. Scores range from 7 to 49. Higher scores indicate poor psychological flexibility.
Change from baseline to immediately after the intervention and 3 month follow-up on the Cognitive Fusion Questionnaire | Change from baseline to immediately after the intervention and 3 month follow-up
  Cognitive Fusion Questionnaire -7 is a 7-item self-report questionnaire measuring cognitive fusion on scale of 1 to 7. Scores range from 7 to 49. Higher scores indicate greater levels of cognitive fusion.
Change from baseline to immediately after the intervention and 3-month follow-up on the Engaged Living Scale | Change from baseline to immediately after the intervention and 3 month follow-up
  Engaged Living Scale -9 is a 9-item self-assessment instrument that measures clarity and engagement with personal values and life fulfillment on a scale of 1 to 5. The total scores range from 9 to 45, and higher scores indicate increased clarity and engagement with personal values and greater life fulfillment.
Change from baseline to immediately after the intervention and 3 month follow-up on the Zarit Burden Interview | Change from baseline to immediately after the intervention and 3 month follow-up
  Zarit Burden Interview is a 12-item self-report questionnaire assessing caregiver burden on a scale of 0 to 4. Higher scores indicate higher levels of burden. The total scores range from 0 to 48, and scores of 17 or greater indicate severe/high burden.

CONTACTS AND LOCATIONS:
Overall Officials: Areum Han, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han A, Oster R, Yuen H, Jenkins J, Hawkins J, Edwards L. Videoconference-Delivered Acceptance and Commitment Therapy for Family Caregivers of People With Dementia: Pilot Randomized Controlled Trial. JMIR Form Res. 2025 Mar 31;9:e67545. doi: 10.2196/67545. PMID 40163859